CLINICAL TRIAL: NCT05278819
Title: Effects of Upper Extremity Elevation and Deep Breathing on Oxygen Saturation and Lung Volume Two to Four Days After Open Heart Surgery
Brief Title: Upper Extremity Elevation and Lungfunction After Open Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael Reinhart (Other)
Collaborators: Region Örebro County (Other); Linkoeping University (Other Government); Örebro University, Sweden (Other)
Responsible Party: Sponsor-Investigator, Michael Reinhart, Physical therapist, Region Örebro County
Organization: Region Örebro County (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 278090
Record Dates: First submitted 2022-02-21; First posted 2022-03-14 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Heart Diseases; Heart Diseases, Ischemic; Heart Disease, Valvular
MeSH Terms: conditions — Heart Diseases; Myocardial Ischemia; Heart Valve Diseases

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- upper extremity elevation (Experimental): performing intervention A (5 repetitions of upper extremity elevation), and then crossed over to intervention B (5 repetitions of upper extremity with deep breathing).
  Interventions: Other: upper extremity elevation; Other: upper extremity elevation with deep breathing
- upper extremity elevation with deep breathing (Experimental): performing intervention B (5 repetitions of upper extremity with deep breathing), and then crossed over to intervention A (5 repetitions of upper extremity elevation).
  Interventions: Other: upper extremity elevation; Other: upper extremity elevation with deep breathing

INTERVENTIONS:
Other: upper extremity elevation — 5 repetitions of active upper extremity elevation in a sitting position
Other: upper extremity elevation with deep breathing — 5 repetitions of active upper extremity elevation with deep breathing in a sitting position

SUMMARY:
The purpose of this study is to assess if arm elevation, with or without simultaneous deep breathing, affects oxygen saturation and lung function on patients two to four days after open heart surgery.

DETAILED DESCRIPTION:
This single center, interventional crossover study will involve patients day 2, 3 or 4 after open heart surgery. Patients who meet the eligibility requirements will be informed about the study and potential risks, given a written informed consent they will be included for intervention being held later on the same day. Randomization will be given to the investigator in a sealed envelope and being opened after base line measurements. Data will then be collected for the randomized intervention and after a wash out period (several minutes) again for the crossover intervention.

ELIGIBILITY:
Inclusion Criteria:

* open heart surgery at university hospital in Örebro

Exclusion Criteria:

* not able to communicate in swedish
* difficulties in cooperating during measurements
* cognitive impairement
* prolonged stay at ICU (still at ICU on the day of investigation)
* ongoing oxygen treatment with more than 5 liter/minut (FiO > 40 %)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-06 (Actual)

PRIMARY OUTCOMES:
peripheral oxygen saturation | 30 minutes

SECONDARY OUTCOMES:
tidal volume | 30 minutes
heart rate | 30 minutes
respiratory rate | 30 minutes
pain - numeric rating scale | 30 minutes
  Pain (sternal, thorax or overall pain) will be measured before and after intervention, NRS will be used (patient rating of perceived pain with a score from 0 to 10)
dyspnea - numeric rating scale | 30 minutes
  Dyspnea will be measured before and after intervention, NRS will be used (patient rating of perceived dyspnea with a score from 0 to 10)
exertion - numeric rating scale | 30 minutes
  exertion will be measured before and after intervention, NRS will be used (patient rating of perceived exertion with a score from 0 to 10)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Örebro, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reinhart M, Jonsson M, Enthoven P, Westerdahl E. Immediate effects of upper limb exercises with and without deep breathing on lung function after cardiac surgery - a randomized crossover trial. J Cardiothorac Surg. 2024 Aug 28;19(1):503. doi: 10.1186/s13019-024-03007-z. PMID 39198875